CLINICAL TRIAL: NCT02325635
Title: A Prospective Randomized Controlled Trial of an Endoscopic Quality Improvement Project-2 (EQUIP-2) to Improve Adenoma Detection in Screening and Surveillance Colonoscopy
Brief Title: A Prospective Trial of an Endoscopic Quality Improvement Project
Acronym: Equip 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GI Quality Improvement Consortium (Other)
Responsible Party: Principal Investigator, Michael Wallace, PI, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 13-002066
Record Dates: First submitted 2014-12-11; First posted 2014-12-25 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Colon Polyps
Keywords: Adenoma Detection; Adenoma Prediction
MeSH Terms: conditions — Colonic Polyps | interventions — Training Support

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training of Endoscopist (Experimental): A series of 1 hour classes with ongoing monitoring and feedback to endoscopist only.
  Interventions: Other: Educational Training
- Deferred Training of Endoscopist (No Intervention): No intervention during the data collection period. Training will be deferred to end of study.

INTERVENTIONS:
Other: Educational Training — Intervention/Training offered to endoscopists only.
  Other Names: Intervention offered to endoscopist only.
  Arms: Training of Endoscopist

SUMMARY:
Randomized prospective multi-site validation study.

DETAILED DESCRIPTION:
GI practice sites that have recently agreed to participate in the GIQuIC program will be randomized on a site-basis, to the EQUIP intervention or control.

Baseline ADR and polyp/surveillance predication accuracy will be collected for approximately 3 months.

Sites randomized to the EQUIP intervention will undergo face-to-face training by a study investigator, followed by active monitoring and feedback.

Control sites will not receive supplemental training and will be monitored by with no feedback. After completion of the study all sites will be offered the intervention (as is standard feedback in GIQuIC ).

ELIGIBILITY:
Inclusion Criteria:

* Endoscopy centers that are new to GIQuIC and have not yet received training
* All endoscopists performing screening and surveillance colonoscopy at the participating center will be invited to participate

Exclusion Criteria:

* Cases that involve acute indications such as bleeding and active colitis will not be included in data pool
* Patients with a family or personal history of a polyposis syndrome or with a personal history of inflammatory bowel disease will also be excluded
* Procedures that are deemed incomplete will be excluded
* Patients with surgically altered anatomy (i.e. prior colectomy) and with poor bowel preparation (Boston bowel preparation score <5, or inadequate to exclude polyps >5mm) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in adenoma detection rates. | 6 months
  The primary outcome will be the change in adenoma detection rates between baseline and the intervention. Validate the effect of a quality improvement training program on the proportion of patients among whom at least one adenoma is detected

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wallace, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Wallace MB, Crook JE, Thomas CS, Staggs E, Parker L, Rex DK. Effect of an endoscopic quality improvement program on adenoma detection rates: a multicenter cluster-randomized controlled trial in a clinical practice setting (EQUIP-3). Gastrointest Endosc. 2017 Mar;85(3):538-545.e4. doi: 10.1016/j.gie.2016.07.042. Epub 2016 Jul 26. PMID 27473182